## **Consent Form**

## <u>Title: Evaluation of the Effects of Virtual Reality Learning Environment on Nursing</u> Student Non-technical Skills Development: A Quasi-Experimental Study

| I hereby consent to participate in the captioned research conducted |
|---|
| by Mr Timothy LAI. |
| I understand that information obtained from this research may be used in future research and |
| published. However, my right to privacy will be retained, i.e. my personal details will not be revealed. |
| The procedure as set out in the attached information sheet has been fully explained. I understand the benefit and risks involved. My participation in the project is voluntary. |
| I acknowledge that I have the right to question any part of the procedure and can withdraw at any |
| time without penalty of any kind. |
| Consent Statement |
| By clicking the button below, you acknowledge that your participation in the study is voluntary, |
| and that you are aware that you may choose to stop participating at any time and for any reason. |
| ☐ Yes. I have read the informed consent information sheet and agree to take part in this |
| research study. |
| Name of Participants: |